CLINICAL TRIAL: NCT05246293
Title: Safety and Tolerability of Tofacitinib in the Treatment of Rheumatoid Arthritis-related Interstitial Lung Disease (RAILDTo Trial).
Brief Title: Tofacitinib in the Treatment of Rheumatoid Arthritis-related Interstitial Lung Disease.
Acronym: RAILDTo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C17-21
Record Dates: First submitted 2022-01-17; First posted 2022-02-18 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-04

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
Keywords: Rheumatoid Arthritis; Interstitial Lung Disease; Usual interstitial pneumonia; Tofacitinib; Rheumatoid Arthritis-related interstitial lung disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: This is a phase 2 open-label study designed to evaluate the safety and tolerability of tofacitinib in RA-ILD patients. Patients who met the inclusion criteria of the study protocol will receive tofacitinib 5 mg BID for 12 months.
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tofacitinib Arm (Experimental): Tofacitinib in doses of 5 mg BID, in RA-ILD patients at stable doses of prednisone ≤ 10 mg/day during the last three months.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib in doses of 5 mg BID, in RA-ILD patients at stable doses of prednisone ≤ 10 mg/day during the last three months.
  Patients who met the inclusion criteria of the study protocol will received tofacitinib 5 mg BID for 12 months

SUMMARY:
Nowadays, no single drug is approved to treat rheumatoid arthritis-related interstitial lung disease (RA-ILD). The medical management of this clinical condition is empirical and controversial. There is preliminary data that tofacitinib may have a beneficial effect in treating RA-ILD. Tofacitinib may have a double role in treating RA-ILD: treat RA disease activity and an anti-fibrotic possible impact. Moreover, tofacitinib may be used as monotherapy for the treatment of rheumatoid arthritis (RA) This is a phase IIa clinical trial to evaluate the safety and tolerability of tofacitinib in RA-ILD patients.

DETAILED DESCRIPTION:
This is a phase 2 open-label study designed to evaluate the safety and tolerability of tofacitinib in RA-ILD patients. Patients who met the inclusion criteria of the study protocol will receive tofacitinib 5 mg BID for 12 months.

Objectives

Primary objectives:

1. To evaluate the safety and tolerability of tofacitinib 5 mg PO BID as monotherapy for managing RA-ILD in RA-ILD patients.
2. To evaluate the pulmonary function of patients treated with tofacitinib PO BID as monotherapy to manage RA-ILD in RA-ILD patients, at baseline, at three months of follow-up, at six months of follow-up, and one year of follow-up.
3. To estimate the efficacy of tofacitinib 5 mg PO BID as monotherapy for the management of RA-ILD, in RA-ILD patients, at three months of follow-up, at six months of follow-up, and at one year of follow-up, according to the ACR 20, 50, 70 response criteria, and the following disease activity scores index: DAS 28, CDAI and SDAI.

All the included patients will receive Tofacitinib in doses of 5 mg BID until the end of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must fulfill ACR/EULAR 2010 RA classification criteria.
2. Patients must have an interstitial lung disease confirmed by a high-resolution computed tomography scan or a surgical lung biopsy. Nonspecific interstitial pneumonia, usual interstitial pneumonia, lymphocytic pneumonia, and organized pneumonia, either by HRCT or surgical biopsy, will be included.
3. Patients must be 18 years of age or older.
4. There is no evidence of active, latent, or inadequately treated infection with Mycobacterium tuberculosis (TB).
5. Patients must discontinue using the non-permitted medications: leflunomide, azathioprine, cyclosporine, tacrolimus, cyclophosphamide, and any biologic disease-modifying drug (bDMDARDs) such as anti-TNF therapy, rituximab, tocilizumab, etc. Patients must have a stable prednisone dose of ≤ 10 mg/ PO/day for at least three months.
6. All patients must have stable doses of prednisone during the last three months of follow-up, and the prednisone dose must be ≤ 10 mg/day. Patients without a prednisone history in the previous three months may also be included in the protocol.

Exclusion Criteria:

1. Seropositivity for the following infections: HIV, HBV, and HCV.
2. Absolute neutrophil count ≤ 1,200/L
3. Absolute platelet count ≤ 100,000 /L
4. Severe renal damage with GFR < 30 ml/min based on CKD-EPI formula.
5. AST or ALT greater than 1.5 times the upper limit of normal AST and ALT levels
6. Severe hepatic, hematologic, gastrointestinal, cardiac, and neurological disease may put the patient´s life at risk regardless of ILD severity.
7. Severe active infections at baseline evaluation, such as pneumonia, urinary tract infections, meningitis.

8 History of drug abuse or alcoholism. 9. History of any malignancy 10. Patients with an FVC < 40% of what is expected will be excluded from the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 52 weeks
  Adverse event: Any untoward medical occurrence in a subject being included in the trial, in which the event may not necessarily have a causal relationship with the treatment. Examples of adverse events are as follows: abnormal test findings, clinically significant symptoms and signs, hypersensitivity reactions, and progression or worsening of RA or RA-ILD.

SECONDARY OUTCOMES:
Forced Vital Capacity (liters) | 52 weeks
  Forced vital capacity (FVC) on spirometry, the data will be presented as percentages of predicted values, according to sex, age, height, and weight.
Carbon monoxide diffusing capacity (DLCO) (mil/min/mmHg) | 52 weeks
  The data will be presented as percentages of predicted values, according to sex, age, height, and weight.
6 minutes walk test | 52 weeks
  walked metters in 6 minutes
Rheumatoid arthritis disease activity according to the simplified disease activity (SDAI) index. | 52 weeks
  The SDAI index consists of the algebraic sum of the following items: tender joint count, swollen joint count, c-reactive protein, rheumatoid arthritis activity according to the patient, disease activity according to the attending physician.
Rheumatoid arthritis disease activity according to the Disease Activity Score Index (DAS28) | 52 weeks
  The DAS28 score is calculated with the tender joint count, swollen joint count, eritrosedimentation rate, patients' global health assesment aacording with the following formula DAS28 = ( 0.56 * sqr(TJC)) + (0.28 * sqr(SJC)) + ( 0.7 * ln(VSG)) + (0.014 * GH)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Rojas-Serrano, MD, PhD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias, Ismael Cosío Villegas
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Ismael Cosío Villegas, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
We will share data, including data dictionaries and analytic code, after presenting the results of the study in a congress or the final publication of the clinical trial. The data will be shared only if a formal research proposal and our local IRB approves this.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after presenting the study results at an international congress or the final publication of the study.
Access Criteria: A formal research proposal, including a research protocol, should be presented to the PI of the study to share the data. The research proposal has to be approved by our local IRB.

REFERENCES:
- [Background] Vacchi C, Manfredi A, Cassone G, Cerri S, Della Casa G, Andrisani D, Salvarani C, Sebastiani M. Tofacitinib for the Treatment of Severe Interstitial Lung Disease Related to Rheumatoid Arthritis. Case Rep Med. 2021 Apr 22;2021:6652845. doi: 10.1155/2021/6652845. eCollection 2021. PMID 33976699
- [Background] Citera G, Mysler E, Madariaga H, Cardiel MH, Castaneda O, Fischer A, Richette P, Chartrand S, Park JK, Strengholt S, Rivas JL, Thorat AV, Girard T, Kwok K, Wang L, Ponce de Leon D. Incidence Rates of Interstitial Lung Disease Events in Tofacitinib-Treated Rheumatoid Arthritis Patients: Post Hoc Analysis From 21 Clinical Trials. J Clin Rheumatol. 2021 Dec 1;27(8):e482-e490. doi: 10.1097/RHU.0000000000001552. PMID 32826657
- [Background] Harigai M. Growing evidence of the safety of JAK inhibitors in patients with rheumatoid arthritis. Rheumatology (Oxford). 2019 Feb 1;58(Suppl 1):i34-i42. doi: 10.1093/rheumatology/key287. PMID 30806708